CLINICAL TRIAL: NCT04891523
Title: Dissecting Probiotic Modulation of Oral Microbiota in Healthy Individuals
Brief Title: Probiotic Modulation of Oral Microbiota
Acronym: PROROBIOTICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Jacques SCHRENZEL (Other)
Responsible Party: Sponsor-Investigator, Prof. Jacques SCHRENZEL, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 320030_197598
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Probiotic (Other): First receive placebo, then active probiotics.
  Interventions: Dietary Supplement: Probiotics-O (Burgerstein); Other: Placebo [inactivated Probiotics-O (Burgerstein)]
- Probiotic-Placebo (Other): First receive active probiotics, then placebo.
  Interventions: Dietary Supplement: Probiotics-O (Burgerstein); Other: Placebo [inactivated Probiotics-O (Burgerstein)]

INTERVENTIONS:
Dietary Supplement: Probiotics-O (Burgerstein) — Topical oral treatment with the probiotic Streptococcus salivarius K12 (BIOTICS-O, Burgerstein) in form of a lozenge, daily, during 3 weeks.
Other: Placebo [inactivated Probiotics-O (Burgerstein)] — Topical oral treatment with the placebo [inactivated probiotic Streptococcus salivarius K12 (BIOTICS-O, Burgerstein)] in form of a lozenge, daily, during 3 weeks.

SUMMARY:
Targeting human microbiota, in particular those of the gastrointestinal tract, by means of prebiotics, probiotics, symbiotics or antibiotics has gained interest for its potential in the management of human health. Oral bacterial communities have been extensively studied over the last decade both in normal and pathological states; however, little data are available on the possibility to modify microbiota composition in a controlled and 'non-aggressive' manner by using probiotics, in order to improve oral health.

Saliva contains microorganisms attached to exfoliated human cells and released from oral biofilms; its microbiota is most similar (proportionally) to those of the dorsal and lateral tongue. In addition, bacteria belonging to genera Porphyromonas, Tannerella and Treponema, which contain species associated with periodontitis, are consistently identified in saliva. Salivary microbial communities are relatively stable and thus potentially interesting as an indicator of oral and general health. Indeed, it has been suggested that interventions aimed at improving oral health should target mucosal microbiota (to which saliva is most similar) in addition to dental microbial communities. Whole saliva also constitutes an alternative to gingival crevicular fluid when analysing analytes present in periodontal pockets. It has been suggested that saliva reflects a consensus inflammatory status of the whole mouth with potentially significant clinical relevance.

Strain K12 of Streptococcus salivarius is available internationally as a food supplement, notably for oral hygiene. Several studies investigated the effectiveness of S. salivarius as a probiotic in the context of pharyngeal infections, halitosis, plaque formation and caries. Our study will focus on the effects of supplementation with this commercially available oral probiotic on the resident microbiota and inflammatory markers in order to identify signatures associated with resistance/susceptibility to colonization by probiotic strains.

DETAILED DESCRIPTION:
OBJECTIVES

This is a monocentric, prospective, cross-over, randomized, double-blinded study in which all participants will receive placebo and active probiotic treatment, 15 of which will first be treated with placebo and then will be given probiotics. The other 15 participants will first get probiotics and then, after a 3-week wash out period, the placebo.

The main objective of the study is to assess changes in salivary microbiota profiles and inflammatory markers following S. salivarius probiotic treatment. Our secondary objective is to identify correlations between specific salivary microbial taxa (subspecies to phylum levels) and inflammatory markers. Clinical outcome is not the focus of this study, although basic information about the oral health will be measured.

METHODOLOGY

BIOTICS-O (Burgerstein) probiotic that will be used is a commercial food supplement available over the counter in the pharmacy as blister packs of 30 lozenges containing 10^9 CFU of S. salivarius K12. Participants will let melt the lozenge after tooth brushing in the evening.

Placebo lozenges (inactivated probiotic) will have the same look, taste and smell as the active treatment lozenges, and they will be administered in the same way as the active treatment lozenges.

Metagenomic analysis of the microbiota:

Indexed paired-end metagenomic libraries will be prepared using DNA extracted from saliva and sequenced for 2x150 cycles on an Illumina NovaSeq 6000 instrument to generate 5-10 million read pairs per sample. Our standard metagenomic analysis pipeline (HUGE-MAP) will be used; it includes: (i) read quality filtering; (ii) removal of replicate sequences; (iii) removal of read pairs that match human genome sequence and, (iv) classification of read pairs with CLARK against the collection of NCBI reference and representative bacterial, archaeal and fungal genomes, as well as Latest RefSeq NCBI genomes of prophages and DNA virus families whose members may infect humans. Functional assignments i.e. profiling the presence/absence and abundance of microbial gene families and pathways will be performed using MG-RAST server. Bacterial abundance will be measured by qPCR and/or relative to the number of reads obtained from the spiked calibrator.

Cytokine measurements:

Salivary cytokines (IL-1β, IL-6, IL-8, TNF-alpha) analysis will be performed using a Salimetrcs Core Cytokine Panel - 4-plex.

OBJECTIVES

This is a monocentric, prospective, cross-over, randomized, double-blinded study in which all participants will receive placebo and active probiotic treatment, 15 of which will first be treated with placebo and then will be given probiotics. The other 15 participants will first get probiotics and then, after a 3-week wash out period, the placebo.

The main objective of the study is to assess changes in salivary microbiota profiles and inflammatory markers following S. salivarius probiotic treatment. Our secondary objective is to identify correlations between specific salivary microbial taxa (subspecies to phylum levels) and inflammatory markers. Clinical outcome is not the focus of this study, although basic information about the oral health will be measured.

METHODOLOGY

BIOTICS-O (Burgerstein) probiotic that will be used is a commercial food supplement available over the counter in the pharmacy as blister packs of 30 lozenges containing 10^9 CFU of S. salivarius K12. Participants will let melt the lozenge after tooth brushing in the evening.

Placebo lozenges (inactivated probiotic) will have the same look, taste and smell as the active treatment lozenges, and they will be administered in the same way as the active treatment lozenges.

Metagenomic analysis of the microbiota:

Indexed paired-end metagenomic libraries will be prepared using DNA extracted from saliva and sequenced for 2x150 cycles on an Illumina NovaSeq 6000 instrument to generate 5-10 million read pairs per sample. Our standard metagenomic analysis pipeline (HUGE-MAP) will be used; it includes: (i) read quality filtering; (ii) removal of replicate sequences; (iii) removal of read pairs that match human genome sequence and, (iv) classification of read pairs with CLARK against the collection of NCBI reference and representative bacterial, archaeal and fungal genomes, as well as Latest RefSeq NCBI genomes of prophages and DNA virus families whose members may infect humans. Functional assignments i.e. profiling the presence/absence and abundance of microbial gene families and pathways will be performed using MG-RAST server. Bacterial abundance will be measured by qPCR and/or relative to the number of reads obtained from the spiked calibrator.

Cytokine measurements:

Salivary cytokines (IL-1β, IL-6, IL-8, TNF-alpha) analysis will be performed using a Salimetrix Core Cytokine Panel - 4-plex..

Samplings will be performed at weeks 1, 4, 7, 10, 13, 16 and 19.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Good oral and general health

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Systemic disease
* Previous enrolment into the current study
* Clinically diagnosed severe oral lesions
* Use of antibiotics and topical oral probiotics within the 3 months preceding the study or during the study
* Dental treatments and use of oral disinfectants within 30 days preceding the study or during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Changes in the overall taxonomic profiles of the salivary bacterial communities (microbiota) following probiotics treatment | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  PERMANOVA test
Changes in the relative abundance of individual bacterial taxa following probiotics treatment | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  ANCOM test
Changes in the absolute abundance of individual bacterial taxa following probiotics treatment | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  Wilcoxon test
Changes in the relative abundance of gene functions following probiotics treatment | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  Wilcoxon test
Changes in the bacterial diversity (Shannon index) | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  Wilcoxon test
Changes in the salivary cytokines levels following probiotics treatment | Will be assessed at the end of a three-week course of no treatment, probiotics or placebo
  Wilcoxon test

SECONDARY OUTCOMES:
Positive and negative correlations between overall bacterial community taxonomic profile and salivary cytokine levels | Will be assessed at weeks 1, 4, 7, 10, 13, 16, 19
  DISTLM
Positive and negative correlations between salivary bacterial taxa and salivary cytokine levels | Will be assessed at weeks 1, 4, 7, 10, 13, 16, 19
  Spearman Rho

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals (HUG), Geneva, Switzerland